CLINICAL TRIAL: NCT00775008
Title: Media Effects Study on Health-Related Content
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Gabrielle Turner-McGrievy, UNC-Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 07-0430-02
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Processing Health Information
Keywords: weight loss, health information, e-health
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- podcast (Experimental)
  Interventions: Behavioral: electronic health information
- Web group (Active Comparator)
  Interventions: Behavioral: electronic health information

INTERVENTIONS:
Behavioral: electronic health information — Participants will receive weight loss information via 1 of 2 different mediums.

SUMMARY:
A media lab study will be conducted to determine the mechanism by which podcasting may exert an effect. This study will examine both physiological (heart rate, skin conductance, etc.) and psychosocial (knowledge, perceived control, elaboration, etc.) measures in participants listening to a podcast on health versus reading health content on the Web. We hypothesize that podcasting will create a greater physiological response than the Web. There will also be more elaboration in the podcasting group. Podcasting will produce greater feelings of control. Changes in knowledge will be greater in the Web group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Be willing to be randomized to either the podcast or Web condition
* Able to attend the intervention session

Exclusion Criteria:

* Not living in the Chapel Hill area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Physiological response | 1 hour

SECONDARY OUTCOMES:
Psychosocial response | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States